CLINICAL TRIAL: NCT01272778
Title: Acute Effect of Four Doses of Lorazepam on Brain Activity Measured by MEG, EEG and the Synchronous Neural Interaction™ Test
Brief Title: Acute Effect of Lorazepam on Brain Activity Measured by Magnetoencephalograpy (MEG) and Electroencephalography (EEG)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orasi Medical, Inc. (Industry)
Responsible Party: Todd Verdoorn, PhD, Chief Scientific Officer, Orasi Medical, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ADE-LDR 10-02
Record Dates: First submitted 2011-01-05; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lorazepam 0.2 mg (Experimental): All subjects receive lorazepam 0.2 mg in this crossover design.
  Interventions: Drug: Lorazepam
- Lorazepam, 0.5 mg (Experimental): All subjects receive lorazepam 0.5 mg in this crossover design.
  Interventions: Drug: Lorazepam
- Lorazepam, 1.0 mg (Experimental): All subjects receive lorazepam 1.0 mg in this crossover design.
  Interventions: Drug: Lorazepam
- Lorazepam, 2.0 mg (Experimental): All subjects receive lorazepam 2.0 mg in this crossover design
  Interventions: Drug: Lorazepam
- Sugar pill (Placebo Comparator): All subjects receive a sugar pill in this crossover design.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorazepam — Oral capsule, 0.2 mg, single acute dose
  Arms: Lorazepam 0.2 mg
Drug: Lorazepam — oral capsule, 0.5 mg, single acute dose
  Arms: Lorazepam, 0.5 mg
Drug: Lorazepam — oral capsule, 1.0 mg, single acute dose
  Arms: Lorazepam, 1.0 mg
Drug: Lorazepam — oral capsule, 2.0 mg, single acute dose
  Arms: Lorazepam, 2.0 mg
Drug: Placebo — oral capsule, single acute dose
  Arms: Sugar pill

SUMMARY:
This placebo-controlled crossover study is intended to measure the effect of four doses of lorazepam on brain activity measured by magnetoencephalography (MEG) and electroencephalography (EEG). This study will conduct MEG and EEG scans as well as simple cognition testing on 16 healthy male volunteers. On each of five study days subjects will be randomized to receive either 0.2, 0.5, 1.0 or 2.0 mg lorazepam or placebo. Brain activity will be measured by MEG and EEG in each subject a total of 4 times each study day: prior to medication administration and 2, 4, and 6 hours after medication administration. Blood samples to determine medication levels and cognition testing will be performed at pre-medication baseline and immediately after each post-medication scan time. Data will be analyzed to identify changes in brain activity compared to baseline and placebo administration using both standard approaches and the Orasi Synchronous Neural Interaction® (SNI) test. This study will test the hypothesis that dose-response changes in brain functional activity can be accurately measured by MEG/EEG in healthy volunteer subjects after single, acute doses of lorazepam.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male between 18 and 35 years of age at the time of screening.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
* Subject is a non-smoker.
* Subject is judged to be in good health based on medical history and brief physical examination and electrocardiogram.
* Subject has normal or corrected to normal visual and auditory acuity.
* Subject agrees to refrain from caffeine 24 hours prior to and then throughout each Study Day.
* Subject agrees to refrain from using alcohol for 48 hours prior to and then throughout each Study Day.

Exclusion Criteria:

* Subject has a diagnosis of a significant neurological condition including Alzheimer's disease, Parkinson's disease, vascular dementia, Lewy body dementia or frontal temporal dementia, human immunodeficiency virus, multiple sclerosis, or severe traumatic brain injury.
* Subject has a history of primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder, delusional disorder) or bipolar disorder.
* Subject has a history of seizures, epilepsy, stroke, peripheral neuropathy, head trauma with persistent post-concussive symptoms, ADHD, dyslexia or other clinically significant neurological disease or cognitive impairment.
* Subject has a lifetime or current history of alcohol or substance abuse/dependence.
* Subject has a history of multiple or severe allergies, or has had an anaphylactic reaction or intolerability to prescription or non-prescription drugs. This includes a documented or subject-verified allergy.
* Subject had an MRI 2 weeks prior to Study Day 2.
* Subject has metal braces or pacemaker that may interfere with the MEG scan.
* Subject is unable to complete the MEG scan procedure.
* The investigator has any concern regarding the safe participation of a subject in the study, or if for any other reason the investigator considers the subject inappropriate for study participation

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Correlated Brain Activity using MEG and SNI analysis | 2 hours after dosing with lorazepam
  The identification and characterization of a pattern of synchronous brain activity that is specifically altered by administration of ascending doses of lorazepam compared to pre-medication baseline and placebo

SECONDARY OUTCOMES:
Correlated Brain Activity using MEG and standard analyses | 2 hours after dosing with lorazepam
  Standard frequency-domain analysis of the MEG data to identify and quantify medication-induced changes in signal power in particular frequency bands associated with brain functional activity

CONTACTS AND LOCATIONS:
Overall Officials: Concetta Forchetti, MD, PhD, Principal Investigator — Alexian Brothers Neurosciences Institute
Locations (1):
- Alexian Brothers Neurosciences Institute, Elk Grove Village, Illinois, United States